CLINICAL TRIAL: NCT00884611
Title: Development of Algorithms for a Hypoglycemic Prevention Alarm
Brief Title: Development of Algorithms for a Hypoglycemic Prevention Alarm: Closed Loop Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-10162008-1321; Stanford eprotocol # 6789 (Other: Stanford University)
Record Dates: First submitted 2009-04-17; First posted 2009-04-21 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Predictive Low Glucose Suspend (Experimental): The pump suspension system consists of the Revel CGM device communicating with a laptop computer that contains the hypoglycemia prediction algorithm. During the 21 night study period, the laptop is placed at the bedside and turned on by the participant at bedtime and off on arising in the morning.The laptop contains a randomization schedule (2:1) that indicats whether the hypoglycemia prediction algorithm will be in operation that night (Predictive Low Glucose Suspend Algorithm ON) or will not be activated (Predictive Low Glucose Suspend Algorithm OFF), to which the participant is blinded.
  Interventions: Device: Predictive Low Glucose Suspend Algorithm ON; Device: Predictive Low Glucose Suspend Algorithm OFF

INTERVENTIONS:
Device: Predictive Low Glucose Suspend Algorithm ON — The algorithm uses a Kalman filter-based model to predict whether the sensor glucose level will fall below 80 mg/dL within a given time period and suspends the insulin pump if this event is predicted.
  Other Names: Intervention Night
Device: Predictive Low Glucose Suspend Algorithm OFF
  Other Names: Control Night

SUMMARY:
This research study, Development of Algorithms for a Hypoglycemic Prevention Alarm, is being conducted at Stanford University Medical Center and the University of Colorado Barbara Davis Center. It is paid for by the Juvenile Diabetes Research Foundation.

The purpose of doing this research study is to understand the best way to stop an insulin infusion pump from delivering insulin to prevent a subject from having hypoglycemia. Nocturnal hypoglycemia is a common problem with type 1 diabetes. This is a pilot study to evaluate the safety of a system consisting of an insulin pump and continuous glucose monitor communicating wirelessly with a bedside computer running an algorithm that temporarily suspends insulin delivery when hypoglycemia is predicted in a home setting.

DETAILED DESCRIPTION:
After the run-in phase, there is a 21-night trial in which each night is randomly assigned 2:1 to have either the predictive low-glucose suspend (PLGS) system active (intervention night) or inactive (control night).

Three predictive algorithm versions were studied sequentially during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older,
2. Type 1 diabetes for at least 1 year
3. Current user of the MiniMed Paradigm Real-Time Revel system and Sof-sensor glucose sensor
4. Hemoglobin A1c level of < 8.0%,
5. Home computer with access to the Internet,
6. At least one CGMglucose value < 70 mg/dL during the most recent 15 nights of CGM glucose data.
7. Not pregnant or planning to become pregnant

Exclusion Criteria:

The exclusion criteria for this study is the following:

1. The presence of a significant medical disorder that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol
2. The presence of any of the following diseases:

   * Asthma if treated with systemic or inhaled corticosteroids in the last 6 months
   * Cystic fibrosis
   * Angina (recurrent heart pain)
   * Past heart attack or coronary artery (heart vessel) disease
   * Past stroke or impairment of blood flow to the brain
   * Other major illness that in the judgment of the investigator might interfere with the completion of the protocol Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment
3. Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
4. Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
5. Severe hypoglycemic event, as described as a seizure, loss of consciousness, severe neurological impairment, or neurological impairment suggestive of hypoglycemia and requiring an emergency department visit or hospitalization within 18 months of enrollment.

Ages: 12 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Buckingham, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Aurora, Colorado

REFERENCES:
- [Result] Buckingham BA, Cameron F, Calhoun P, Maahs DM, Wilson DM, Chase HP, Bequette BW, Lum J, Sibayan J, Beck RW, Kollman C. Outpatient safety assessment of an in-home predictive low-glucose suspend system with type 1 diabetes subjects at elevated risk of nocturnal hypoglycemia. Diabetes Technol Ther. 2013 Aug;15(8):622-7. doi: 10.1089/dia.2013.0040. Epub 2013 Jul 24. PMID 23883408

RESULTS

PARTICIPANT FLOW:
Groups:
- Predictive Suspend: Participants had continuous glucose monitoring (CGM) using a glucose sensor and received insulin from an insulin pump during sleep. On intervention nights, participants received insulin uising an algorithm that allowed a computer to assess the data received from the CGM sensor and suspend insulin delivery to avoid potential hypoglycaemia. On control night, participants received insulin delivery as normally received by the insulin pump. Participants had 2 intervention nights to each control night.
Period: Overall Study
Arm/Group | Predictive Suspend
Started | 20
Enrolled, Not Treated | 1
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Predictive Suspend
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Nights With CGM (Continuous Glucose Monitor) Sensor Values < 60 mg/dL
Description: Nights with CGM sensor values < 60 mg/dL were considered to be undesirable. A Kalman filter-based model algorithm predicted whether the sensor glucose level would fall below 80 mg/dL and would suspend insulin delivery as needed. Participants may have received treatment using one or more of the following algorithms: Algorithm 1 had a hypoglycaemic prediction horizon of 70 minutes; algorithm 2: 50 minutes; algorithm 3: 30 minutes.
Time Frame: 21 days
Population: Participants who were treated and had data for the respective algorithm were included in the analysis.
Measure: Number; unit: percentage of nights
Units Other Than Participants: Nights
Groups:
- Algorithm 1 - Control Nights; Algorithm 1 - Intervention Nights: Algorithm 1 had a hypoglycaemic prediction horizon of 70 minutes.
  Participants had continuous glucose monitoring (CGM) using a glucose sensor and received insulin from an insulin pump during sleep. On intervention nights, participants received insulin uising an algorithm that allowed a computer to assess the data received from the CGM sensor and suspend insulin delivery to avoid potential hypoglycaemia. On control night, participants received insulin delivery as normally received by the insulin pump. Participants had 2 intervention nights to each control night.
- Algorithm 2 - Control Nights; Algorithm 2 - Intervention Nights: Algorithm 2 had a hypoglycaemic prediction horizon of 50 minutes.
  Participants had continuous glucose monitoring (CGM) using a glucose sensor and received insulin from an insulin pump during sleep. On intervention nights, participants received insulin uising an algorithm that allowed a computer to assess the data received from the CGM sensor and suspend insulin delivery to avoid potential hypoglycaemia. On control night, participants received insulin delivery as normally received by the insulin pump. Participants had 2 intervention nights to each control night.
- Algorithm 3 - Control Nights; Algorithm 3 - Intervention Nights: Algorithm 3 had a hypoglycaemic prediction horizon of 30 minutes.
  Participants had continuous glucose monitoring (CGM) using a glucose sensor and received insulin from an insulin pump during sleep. On intervention nights, participants received insulin uising an algorithm that allowed a computer to assess the data received from the CGM sensor and suspend insulin delivery to avoid potential hypoglycaemia. On control night, participants received insulin delivery as normally received by the insulin pump. Participants had 2 intervention nights to each control night.
Arm/Group | Algorithm 1 - Control Nights | Algorithm 1 - Intervention Nights | Algorithm 2 - Control Nights | Algorithm 2 - Intervention Nights | Algorithm 3 - Control Nights | Algorithm 3 - Intervention Nights
Number analyzed (Participants) | 5 | 5 | 12 | 12 | 9 | 9
Number analyzed (Nights) | 38 | 67 | 48 | 108 | 37 | 77
percentage of nights | 24 | 12 | 25 | 11 | 22 | 8

2. Secondary Outcome: Percentage of Nights With CGM Values >180 mg/dL
Description: Nights with CGM sensor values >180 mg/dL were considered to be undesirable. Participants may have received treatment using one or more of the following algorithms: Algorithm 1 had a hypoglycaemic prediction horizon of 70 minutes; algorithm 2: 50 minutes; algorithm 3: 30 minutes.
Time Frame: 21 days
Population: Participants who were treated and had data for the respective algorithm were included in the analysis.
Measure: Number; unit: percentage of nights
Units Other Than Participants: Nights
Arm/Group | Algorithm 1 - Control Nights | Algorithm 1 - Intervention Nights | Algorithm 2 - Control Nights | Algorithm 2 - Intervention Nights | Algorithm 3 - Control Nights | Algorithm 3 - Intervention Nights
Number analyzed (Participants) | 5 | 5 | 12 | 12 | 9 | 9
Number analyzed (Nights) | 38 | 67 | 48 | 108 | 37 | 77
percentage of nights | 63 | 78 | 29 | 56 | 49 | 60

3. Secondary Outcome: Mean Morning Blood Glucose (BG)
Description: Desirable glucose level was 70-180 mg/mL. Average of all morning BG data is presented. Participants may have received treatment using one or more of the following algorithms: Algorithm 1 had a hypoglycaemic prediction horizon of 70 minutes; algorithm 2: 50 minutes; algorithm 3: 30 minutes.
Time Frame: 21 days
Population: Participants who were treated and had data for the respective algorithm were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Algorithm 1 - Control Nights | Algorithm 1 - Intervention Nights | Algorithm 2 - Control Nights | Algorithm 2 - Intervention Nights | Algorithm 3 - Control Nights | Algorithm 3 - Intervention Nights
Number analyzed (Participants) | 5 | 5 | 12 | 12 | 9 | 9
mg/dL | 125 (53) | 158 (52) | 138 (63) | 151 (57) | 133 (57) | 144 (48)

ADVERSE EVENTS:
Time Frame: 21 days
Description: Only treated participants were evaluable for adverse events.
Groups:
- Control Night (PLGS Algorithm OFF): Participants had continuous glucose monitoring (CGM) using a glucose sensor and received insulin from an insulin pump during sleep. On intervention nights, participants received insulin uising an algorithm that allowed a computer to assess the data received from the CGM sensor and suspend insulin delivery to avoid potential hypoglycaemia. On control night, participants received insulin delivery as normally received by the insulin pump. Participants had 2 intervention nights to each control night.
  Data for control night are reported in this group.
- Intervention Night (PLGS Algorithm ON): Participants had continuous glucose monitoring (CGM) using a glucose sensor and received insulin from an insulin pump during sleep. On intervention nights, participants received insulin uising an algorithm that allowed a computer to assess the data received from the CGM sensor and suspend insulin delivery to avoid potential hypoglycaemia. On control night, participants received insulin delivery as normally received by the insulin pump. Participants had 2 intervention nights to each control night.
  Data for intervention nights are reported in this group.
Arm/Group | Control Night (PLGS Algorithm OFF) | Intervention Night (PLGS Algorithm ON)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No